CLINICAL TRIAL: NCT02617056
Title: Objective Assessment of Behavioral Associations of Patients With Dementia
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: N1932-P; RX001932-01 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Psychomotor Agitation
Keywords: electrodermal response
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational group: Subjects with dementia

SUMMARY:
It is generally acknowledged that patients with dementia are best cared for at home. However, outbursts of various behavioral disturbances, e.g., combativeness, appear in most cases and often necessitate institutionalization. These outbursts are often without apparent warning, which limits preventive interventions. The measurement of the electrical activity of the skin is well-studied as an indicator of stress or agitation. The investigators propose to monitor the electrical activity of skin in patients with dementia in order to determine whether any sign of agitation may occur before the outburst. If skin electrical activity gives sufficient warning, then preventive interventions may be tried. If successful, the ability to predict and prevent outbursts of behavioral disturbances will allow patients to be cared for at home for longer periods. It is the primary aim of this project to determine whether skin electrical activity gives such a warning; possible preventive measures will be the subject of future studies.

DETAILED DESCRIPTION:
1. Objective(s): The key goal of this project is to develop methods for objectively monitoring and, ultimately, predicting outbursts of aberrant behaviors commonly seen among patients with a variety of neuropsychiatric conditions: dementia, PTSD, TBI, and schizophrenia. This initial study will be on patients with dementia. The analytic focus is on the measurement of electrodermal activity (EDA), a widely-studied physiological recording that indicates sympathetic tone; the central hypothesis in this approach is that sympathetic tone will increase prior to an outburst and, therefore, may allow therapeutic interventions to prevent it. Alterations of sympathetic activity have been implicated in the literature for each of these four conditions. Here, EDA recording holds the advantages of requiring neither effort nor communication on the part of the subject, and of being a noninvasive procedure. These factors make EDA potentially useful for the clinical assessment of arousal among patients with dementia, which will be the first of the specific groups studied under this protocol.
2. Research Design: The general design of all of these studies is the monitoring of EDA in subjects with a small device that can be worn on the wrist, ankle or arm; patterns of spontaneous EDA will then be assessed for features that may predict the occurrence of an outburst. In the initial study of dementia patients, the investigators will first survey EDA responses in commonly used paradigms (e.g., visual stimulus, EDA response). Currently, little is known about EDA in this population, and the investigators redress this by (1) establishing behavioral and physiological baselines for each subject in the study, (2) determining how these two classes of dependent measures cohere, and (3) evaluating whether patterns of EDA differ as a function of aberrant behaviors that are often seen in dementia: wandering, combativeness, and "sundowning" (agitation that typically develops late in the day). These behaviors are often grouped in the literature under the term "disorders of arousal", and are clinically well known to present as signs of disorientation and in some cases, distress. (4) Moreover, quantitative assessment of EDA change conceivably may reveal patterns that may signal the onset of problem behaviors.

   Each subject will serve as his/her own control, providing within-subject measures of EDA signal over time and its correlation with aberrant behaviors. It is worth noting that the key EDA measures are not subject to bias based on experimenter ratings. Further, the aberrant behaviors will also be rated over time, using quantitative rating scales for each of them. In a second class of analyses, the investigators will perform group contrasts of subjects with and without these aberrant behaviors, as operationally defined by rating scales, to determine if patients with these problem behaviors are distinctive as a group with respect to EDA patterns. All statistical analysis will be performed on anonymized data, blind to group membership.
3. Methodology: EDA will be measured by standard techniques in all subjects: electrodes may be placed on the hands, feet, ankles, wrists, or arm according to preference and configured to measure conductivity or potential. In one portion of the study, a wearable device to measure EDA will be used to determine whether EDA predicts the occurrence of an outburst. In the study with dementia patients, assessments will be performed at an inpatient dementia care facility at the Bedford VAMC (GRECC). Over a two-year period, the investigators anticipate enrolling 60 subjects. Recruitment criteria include toleration of the EDA recording device worn on the wrist (similar to a watch) or the ankle. Skin potential, skin conductance, and membrane electrical power will be monitored and data recorded electronically. Data will be de-identified by assigning the serial subject number to each patient; a table linking the number to the subject's identity will be kept on a secure VA server, allowing re-identification after data analysis.
4. Findings: If successful, EDA may predict an outburst of aberrant behavior with enough lead time to permit a preventive intervention.
5. Clinical Relationships: The investigators hypothesize that: (a) stable physiologic baselines can be obtained for EDA measures, (b) EDA signals are altered as a function of aberrant behaviors ("disorders of arousal") on a within-subject basis, and (c) group differences will emerge between samples of patients with and without these aberrant behaviors.
6. Impact/Significance: If the EDA were borne out as a sensitive measure of disorders of arousal, this measure may find application in the assessment and treatment of dementia.

ELIGIBILITY:
Inclusion Criteria:

* any patient admitted to dementia unit at Bedford VAMC

Exclusion Criteria:

* inability to cooperate with electrodermal measurements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients in dementia unit have advanced dementia; a small number of young adult controls will be studied to validate electrodermal measurements
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Electrodermal activity | Continuously over a period of 4-6 hours
  The purpose of this trial is to determine whether a signal of electrodermal activity (EDA) will precede an outburst of a behavioral disturbance by enough time to permit an intervention to prevent that behavior. This is a pilot project to test this hypothesis; subsequent studies will test the effectiveness of interventions. Therefore, the primary outcome sought is the detection of such a signal. EDA includes skin potential and skin conductivity. The time course of these two measurements form electrical signals. The shape of these signals will be characterized by mean value, spectral analysis and principle component analysis. The three analyses of two signals lead to six categories of information about the subject that will be examined as predictors of an outburst. Each subject will serve as his own control. More specifically, a successful outcome of this pilot project is that information from these six categories, alone or in combination, can predict an outburst.

SECONDARY OUTCOMES:
Association of behaviors with electrodermal activity | Continuously over a period of 4-6 hours
  While observing a subject to detect a signal for measure 1 above, we expect to detect minor variations of electrodermal activity that may correlate with objects in the environment, indicating a stress response that may not be apparent from the subject's demeanor. This may reveal unsuspected stress factors in the environment, the reduction of which may improve the subject's well being.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greco, MD PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request after publication.

REFERENCES:
- [Background] Greco FA, Deutsch CK. Carl Gustav Jung and the psychobiology of schizophrenia. Brain. 2017 Jan;140(1):e1. doi: 10.1093/brain/aww273. Epub 2016 Nov 15. No abstract available. PMID 28031224
- [Result] Deutsch CK, Patnaik PP, Greco FA. Is There a Characteristic Autonomic Response During Outbursts of Combative Behavior in Dementia Patients? J Alzheimers Dis Rep. 2021 May 4;5(1):389-394. doi: 10.3233/ADR-210007. PMID 34189410